CLINICAL TRIAL: NCT03334526
Title: Corticospinal and Neuromuscular Plasticity Induced by Real and Imaginary Contractions.
Brief Title: Study of the Reaction of the Brain to Various Stimulations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GREMEAUX 2017
Record Dates: First submitted 2017-10-13; First posted 2017-11-07 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Corticospinal Plasticity; Neuromuscular Plasticity
MeSH Terms: interventions — Physical Conditioning, Human; Electric Stimulation

STUDY DESIGN:
Intervention Model Description: this study is interventional because of it acts on the physical and respiratory capacities of patients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- healthy volunteers (Experimental)
  Interventions: Other: physical training; Other: mental training; Other: electrical stimulation

INTERVENTIONS:
Other: physical training — workout on treadmill requiring the muscles of the lower limbs mostly in concentric (ascent) or eccentric (downhill)
Other: mental training — The task to imagine for the training group will be an abduction of the thumb
Other: electrical stimulation — electrical stimulation of the muscles

SUMMARY:
Physical activity is considered a therapeutic strategy in its own right in a vast majority of disabling chronic disorders. It leads to an increase in physical and probably cognitive capacity, thanks to its effects on both metabolism (muscle hypertrophy, improvement in oxidative metabolism) and the nervous system (neuroplasticity). Nonetheless, even though there is a consensus on the positive effects of physical exercise (PE) on cerebral plasticity, the physiological mechanisms by which PE affects neuroplasticity, in particular depending on the mode of muscle contraction, are still hypothetical. Moreover, several recent studies have shown that mental learning (ML) by motor imagery improves motor performance, thus making it of interest in a context of rehabilitation, in particular in situations where PE is transient of definitively impossible. Yet, the mechanisms and brain structures involved in motor learning by ML have not been established so far. Finally, on the basis of clinical observations concerning the key role of sensory input in motor function, the hypothesis that increased demand on this input by electrical stimulation (ES) as a means to improve motor function has been proposed. However, the mechanisms by which this type of stimulation could induce neuroplasticity is still to be elucidated.

ELIGIBILITY:
Inclusion Criteria:

* persons who have provided written consent
* healthy subjects
* national health insurance cover
* age 18 to 60 years

Exclusion Criteria:

* personal or family history of epilepsy
* pacemakers or other apparatus likely to interfere with the magnetic field
* history of psychiatric disease
* Persons under guardianship or wards of court
* Pregnant or breast-feeding women
* problem perceived during the neurological examination which could bias the results of the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 174 (Actual)
Dates: Start 2017-11-09 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

PRIMARY OUTCOMES:
level of corticospinal excitability | through study completion, an average of 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Dupont W, Papaxanthis C, Lebon F, Madden-Lombardi C. Mental Simulations and Action Language Are Impaired in Individuals with Aphantasia. J Cogn Neurosci. 2024 Feb 1;36(2):261-271. doi: 10.1162/jocn_a_02084. PMID 37944123